CLINICAL TRIAL: NCT06257446
Title: The Influence of Mesolimbic-hippocampal Interactions on Episodic Memory During Active Information Seeking
Brief Title: InformationSeekingMesolimbicEngagementStudy1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R01DA055259-1; R01DA055259 (NIH)
Record Dates: First submitted 2024-01-31; First posted 2024-02-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Motivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motivation (Experimental): Trials in which participants are motivated by agency or not in a within-subjects design
  Interventions: Behavioral: Task Instructions

INTERVENTIONS:
Behavioral: Task Instructions — Participants will be given cued instructions as to whether they are in a high or low motivation condition

SUMMARY:
Study 1 will use a novel Game Show task, in which the investigators manipulate participant's agency to control their learning environment to specify unguided exploration.

DETAILED DESCRIPTION:
Study 1 will use a novel Game Show task, in which the investigators manipulate participant's agency to control their learning environment to specify unguided exploration. In the encoding session, participants play the producer for a game show. On each trial, participants are shown a trial-unique contestant (2s), and then they select one of 3 presented doors to reveal a hidden object (4 seconds). The selected door is then highlighted (2-4s), which is then removed to show a trial-unique object image, which is framed as a prize (2s). On exploration trials, participants actively select which door to open. On control trials, the participant is forced to select a highlighted door, fostering passive rather than active information seeking. Unbeknownst to participants, there is no relationship between selected doors and revealed objects, as objects are pre-selected for each trial. Thus, timing, motor demands, and visual information are fixed across conditions. Participants will complete 3 runs of both the exploration and control condition, with each run containing 20 trials. Temporal jitters are placed between cues and outcomes and between trials, as determined by design optimization software77. Run will be pseudo-randomized across participants so no more than 2 runs of the same condition will appear in a row. Following encoding, participants will complete immediate and delayed item-associative memory test. On each trial of the memory test, participants will view the characters presented during exploration and control trials as well as new foil characters. If a participant indicates that they have previously seen a character before, the participants will be shown three object images encountered during encoding, and decide which item served as a prize for that specific character. In this way, the investigators can resolve memory for contestants (i.e., cues), and associative binding across contestants and prizes (i.e., cue-outcome). Participants memory will be tested for half the stimuli immediately and at a 24-hour delay.

ELIGIBILITY:
Inclusion Criteria:

* 20/40 far acuity (either corrected or uncorrected)
* In good medical health

Exclusion Criteria:

* History of head injury
* History of illness with Central Nervous Systems implications
* On Medications that Affect blood flow response and alertness
* Consumption of smoking and/or coffee 30 minutes prior to laboratory testing
* Placement of a device contraindicated for magnetic resonance imaging including cardia pacemaker, aneurysm clip, cochlear implants, pregnancy, intra-uterine device, shrapnel, metal fragments in the eyes, neurostimulators
* Weight > 250lbs
* Claustrophobia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Mesolimbic-hippocampal Interactions | During Procedure
  Functional Magnetic Resonance Imaging Activation characterizing mesolimbic-hippocampal interactions
Episodic Memory | 24-hours after Procedure
  Item and Associative memory for memoranda shown during the task

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared on the open science framework.
Supporting Information: Analytic Code
Time Frame: Data will be shared within 1 year of study completion, and it will be available for at least 10 years.